CLINICAL TRIAL: NCT03766880
Title: MR-based Models for Noninvasive Detection of Clinically Significant Portal Hypertension in Cirrhosis (CHESS1802)
Brief Title: MR-based Models for Clinically Significant Portal Hypertension in Cirrhosis (CHESS1802)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Zhongda Hospital (Other); Beijing 302 Hospital (Other); Affiliated Lishui Hospital of Zhejiang University (Unknown); Shandong Provincial Hospital (Other Government); Xingtai People's Hospital (Other); The First Hospital of Zhengzhou University (Unknown); Shanghai Public Health Clinical Center, Fudan University (Unknown); LanZhou University (Other); Southern Medical University, China (Other); Ankara University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Hepatic Hemodynamic Lab, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHESS1802
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hypertension, Portal
Keywords: clinically significant portal hypertension, hepatic venous pressure gradient, MR imaging
MeSH Terms: conditions — Hypertension, Portal | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Participants will receive MR imaging, transjugular HVPG measurement, and analysis per protocol.
  Interventions: Procedure: Transjugular HVPG measurement; Procedure: MR imaging

INTERVENTIONS:
Procedure: Transjugular HVPG measurement — By means of catheterization of a hepatic vein with a balloon catheter.
Procedure: MR imaging — MR images for the post-processing analysis

SUMMARY:
Clinically significant portal hypertension (CSPH) is associated with an incremental risk of esophageal varices and overt clinical decompensations in cirrhosis. However, hepatic venous pressure gradient (HVPG) measurement, the gold standard for defining CSPH (HVPG≥ 10mmHg) is invasive and therefore not suitable for routine clinical practice.

This is a multi-center diagnostic trial conducted at high-volume liver centres designed to determine the accuracy of MR-based models (investigational technology) for noninvasive detection of a CSPH in patients with cirrhosis. Transjugular HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH.

DETAILED DESCRIPTION:
Clinically significant portal hypertension (CSPH) is associated with an incremental risk of esophageal varices and overt clinical decompensations in cirrhosis. However, hepatic venous pressure gradient (HVPG) measurement, the gold standard for defining CSPH (HVPG≥ 10mmHg) is invasive and therefore not suitable for routine clinical practice.

This is a multi-center diagnostic trial conducted at high-volume liver centres (Zhongda Hospital, Medical School of Southeast University; Affiliated Lishui Hospital of Zhejiang University; Shandong Provincial Hospital affiliated to Shandong University; Beijing 302 Hospital; Xingtai People's Hospital; Shunde Hospital, Southern Medical University; The First Hospital of Zhengzhou University; Shanghai Public Health Clinical Center, Fudan University; The First Hospital of Lanzhou University; Nanfang Hospital of Southern Medical University; Ankara University School of Medicine) designed to determine the accuracy of MR-based models (investigational technology) for noninvasive detection of a CSPH in patients with cirrhosis. Transjugular HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* With written informed consent
* Confirmed liver cirrhosis based on liver biopsy or clinical findings
* Scheduled to undergo clinically-indicated transjugular HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter
* Has undergone> MR imaging within 14 days to hepatic vein catheterization
* No hepatic-portal vein interventional therapy between MR imaging and hepatic vein catheterization

Exclusion Criteria:

* A contraindication to MR imaging, in particular pacemakers or implantable defibrillators, cochlear implants, neurosurgical clips, intra-orbital or brain metallic foreign bodies, endo prothesis since less than 4 weeks or osteosynthesis material since less than 6 weeks
* Unable to comply with breathing or other imaging related instructions resulting in inability to obtain diagnostic quality MR imaging studies
* Contraindication to the injection of contrast agent: pregnancy, lactation, history of allergic reaction to contrast agent injection.
* Prior transjugular intrahepatic portosystem stent-shunt surgery
* Prior devascularization operation
* Has received a liver transplant
* Any active, serious, life-threatening disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance of MR-based Models | 1 day
  Accuracy, sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of MR-based models for noninvasive detection of CSPH when compared to HVPG as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, MD, Principal Investigator — Nanfang Hospital, Southern Medical University; Shenghong Ju, MD, Principal Investigator — Zhongda Hospital
Locations (11):
- China (10):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shunde Hospital, Southern Medical University, Shunde, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongda Hospital, Medical School of Southeast University, Nanjing, Jiangsu
  - Shandong Provincial Hospital affiliated to Shandong University, Jinan, Shandong
  - Shanghai Public Health Clinical Center, Fudan University, Shanghai, Shanghai Municipality
  - Affiliated Lishui Hospital of Zhejiang University, Lishui, Zhejiang
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Sun R, Limkin EJ, Vakalopoulou M, Dercle L, Champiat S, Han SR, Verlingue L, Brandao D, Lancia A, Ammari S, Hollebecque A, Scoazec JY, Marabelle A, Massard C, Soria JC, Robert C, Paragios N, Deutsch E, Ferte C. A radiomics approach to assess tumour-infiltrating CD8 cells and response to anti-PD-1 or anti-PD-L1 immunotherapy: an imaging biomarker, retrospective multicohort study. Lancet Oncol. 2018 Sep;19(9):1180-1191. doi: 10.1016/S1470-2045(18)30413-3. Epub 2018 Aug 14. PMID 30120041
- [Background] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833
- [Background] Wang K, Lu X, Zhou H, Gao Y, Zheng J, Tong M, Wu C, Liu C, Huang L, Jiang T, Meng F, Lu Y, Ai H, Xie XY, Yin LP, Liang P, Tian J, Zheng R. Deep learning Radiomics of shear wave elastography significantly improved diagnostic performance for assessing liver fibrosis in chronic hepatitis B: a prospective multicentre study. Gut. 2019 Apr;68(4):729-741. doi: 10.1136/gutjnl-2018-316204. Epub 2018 May 5. PMID 29730602
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Lambin P, Leijenaar RTH, Deist TM, Peerlings J, de Jong EEC, van Timmeren J, Sanduleanu S, Larue RTHM, Even AJG, Jochems A, van Wijk Y, Woodruff H, van Soest J, Lustberg T, Roelofs E, van Elmpt W, Dekker A, Mottaghy FM, Wildberger JE, Walsh S. Radiomics: the bridge between medical imaging and personalized medicine. Nat Rev Clin Oncol. 2017 Dec;14(12):749-762. doi: 10.1038/nrclinonc.2017.141. Epub 2017 Oct 4. PMID 28975929
- [Derived] Wang C, Huang Y, Liu C, Liu F, Hu X, Kuang X, An W, Liu C, Liu Y, Liu S, He R, Wang H, Qi X. Diagnosis of Clinically Significant Portal Hypertension Using CT- and MRI-based Vascular Model. Radiology. 2023 Apr;307(2):e221648. doi: 10.1148/radiol.221648. Epub 2023 Jan 31. PMID 36719293
- [Derived] Liu Y, Tang T, Ormeci N, Huang Y, Wang J, Li X, Li Z, An W, Liu D, Zhang C, Liu C, Liu J, Liu C, Wang G, Mosconi C, Cappelli A, Bruno A, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Ellik Z, Asiller OO, Li L, Zhang H, Kang N, Xu D, He R, Wang Y, Bu Y, Gu Y, Ju S, Golfieri R, Qi X. Noncontrast-enhanced MRI-based Noninvasive Score for Portal Hypertension (CHESS1802): An International Multicenter Study. J Clin Transl Hepatol. 2021 Dec 28;9(6):818-827. doi: 10.14218/JCTH.2021.00177. Epub 2021 Sep 30. PMID 34966645
- [Derived] Liu Y, Ning Z, Ormeci N, An W, Yu Q, Han K, Huang Y, Liu D, Liu F, Li Z, Ding H, Luo H, Zuo C, Liu C, Wang J, Zhang C, Ji J, Wang W, Wang Z, Wang W, Yuan M, Li L, Zhao Z, Wang G, Li M, Liu Q, Lei J, Liu C, Tang T, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Ellik Z, Asiller OO, Liu Z, Teng G, Chen Y, Hou J, Li X, He X, Dong J, Tian J, Liang P, Ju S, Zhang Y, Qi X. Deep Convolutional Neural Network-Aided Detection of Portal Hypertension in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2998-3007.e5. doi: 10.1016/j.cgh.2020.03.034. Epub 2020 Mar 21. PMID 32205218